CLINICAL TRIAL: NCT07235722
Title: Exploring Resilience. A Qualitative Study of an Intervention After Intimate Partner Violence.
Brief Title: How a Resilience-Focused Intervention is Perceived by Women Subjected to Domestic Violence
Acronym: EMBER-2
Status: Not yet recruiting | Type: Observational
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Other Study IDs: EMBER-2; 2025-04335-01 (Other: Swedish Ethical Review Authority)
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Shame; Intimate Partner Violence; Domestic Violence Exposure; Resilience, Psychological
Keywords: Qualitative; interview; Intimate Partner Violence; Domestic Violence; domestic violence exposure; gender-based violence; Shame; Resilience, Psychological

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EMBER-intervention participants: Women subjected to intimate partner violence at the NCK outpatient clinic
  Interventions: Behavioral: Qualitative interview

INTERVENTIONS:
Behavioral: Qualitative interview — A semi-structured interview

SUMMARY:
At Uppsala University Hospital, there is an outpatient clinic for women subjected to intimate partner violence. In order to explore how patients experience the biopsychosocial resilience-based intervention in use at the clinic and how well the intervention fits the needs of the patients, 30 patients from different stages of their contact at the clinic and with diverse life situations and background are enrolled. The researchers will carry out individual in-person interviews, each lasting approximately 60 minutes, based on a semi-structured set of questions. The questions concern the participant´s life situation, resilience and self-perceived needs, how well the intervention has met those needs and how it was perceived by the participant. The interviews are audio-recorded and transcribed verbatim for thematic analysis.

ELIGIBILITY:
Inclusion Criteria:

* Enrolled in the EMBER intervention at the NCK outpatient clinic.

Exclusion Criteria:

* Any situation that, in the opinion of the Investigator, would compromise the safety of the patient or the quality of the data.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The participants are patients at the NCK outpatient clinic at Uppsala University Hospital, due to experiences of being subjected to intimate partner violence. Due to clinic admission criteria, the population is limited to women over 18 of age. Participants are enrolled by strategic sampling to assure a diverse sample across variables of health, age, ethnicity, socio-economy and time enrolled at the clinic.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Patient experiences of EMBER | To be conducted at the time of enrollment
  Interview questions exploring experiences and attitudes regarding the EMBER intervention

SECONDARY OUTCOMES:
Needs and resilience | to be conducted at the time of enrollment
  Interview questions concerning perceptions and beliefs regarding what is needed for recovery after intimate partner violence

IPD SHARING:
Plan to Share IPD: No